CLINICAL TRIAL: NCT00915798
Title: Smoking, Neurocircuitry and Genes in Adult ADHD
Brief Title: Association Between Smoking, Brain Activity, Genes, and ADHD
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jean Gehricke, Associate Professor, University of California, Irvine
Other Study IDs: HS 2009-6740; K01DA025131 (NIH)
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Smoking; Withdrawal Nicotine; ADHD
MeSH Terms: conditions — Smoking; Attention Deficit Disorder with Hyperactivity | interventions — Natural Family Planning Methods

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Blood samples for genotyping
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Smokers with ADHD: Smokers with ADHD participated in one overnight abstinence condition (withdrawal) and one smoking condition (smoking the first cigarette of the morning).
  Interventions: Behavioral: Cigarette smoking; Behavioral: Abstinence
- Nonsmokers with ADHD: Nonsmokers with ADHD participated in one condition.
  Interventions: Behavioral: Abstinence
- Control smokers: Control smokers participated in one overnight abstinence condition (withdrawal) and one smoking condition (smoking the first cigarette of the morning).
  Interventions: Behavioral: Cigarette smoking; Behavioral: Abstinence
- Control nonsmokers: Control nonsmokers participated in one condition.
  Interventions: Behavioral: Abstinence

INTERVENTIONS:
Behavioral: Cigarette smoking — Participants had an fMRI scan during an experimental task consisting of mathematical problems after smoking a cigarette.
  Groups: Control smokers; Smokers with ADHD
Behavioral: Abstinence — Participants had an fMRI scan during an experimental task consisting of mathematical problems after smoking abstinence.

SUMMARY:
The study investigated the underlying mechanisms of smoking in young adults by examining the associations between smoking, brain activity, dopamine genes, and attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The study investigated the underlying mechanisms of smoking in young adults by examining the associations between smoking, brain activity, dopamine genes, and attention deficit hyperactivity disorder (ADHD). Four groups of young adults were recruited: (1) smokers with ADHD; (2) nonsmokers with ADHD; (3) normative control smokers; and (4) normative control nonsmokers. Smoking was assessed via questionnaires and salivary cotinine levels. Brain activity was examined via functional Magnetic Resonance Imaging (fMRI). Each nonsmoker underwent an fMRI scan during an experimental task consisting of mathematical problems. Smokers underwent two fMRI scans during similar experimental tasks under the following two conditions: (1) after smoking a cigarette and (2) after overnight abstinence. The association between the DRD4-7 repeat allele and smoking was explored.

ELIGIBILITY:
Inclusion Criteria:

1. Smokers with ADHD

   * Cigarette smoking for the last year
   * ADHD diagnosis
2. Nonsmokers with ADHD

   * No history of regularly smoking cigarettes
   * ADHD diagnosis
3. Normative control smokers

   * Cigarette smoking for the last year
   * No history and diagnosis of ADHD
4. Normative control nonsmokers

   * No history of regularly smoking cigarettes
   * No history and diagnosis of ADHD

Exclusion Criteria:

* Children under the age of 18
* Adults above the age of 45
* Pregnancy or planning to become pregnant
* Any major medical illness
* Any mental disorders that require medication (except stimulant medication)
* Any contraindications to fMRI scanning
* Not speaking English

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Commuity sample
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2009-07; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-G. Gehricke, Ph.D., M.A., Principal Investigator — University of California, Irvine
Locations (1):
- 2500 Red Hill Avenue, Santa Ana, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gehricke JG, Swanson JM, Duong S, Nguyen J, Wigal TL, Fallon J, Caburian C, Muftuler LT, Moyzis RK. Increased brain activity to unpleasant stimuli in individuals with the 7R allele of the DRD4 gene. Psychiatry Res. 2015 Jan 30;231(1):58-63. doi: 10.1016/j.pscychresns.2014.10.021. Epub 2014 Nov 4. PMID 25481571
- [Derived] Gehricke JG, Gevorkian J, Stehli A, Alejo SD, Dawson M, Kopelevich A. Discrepancies in the Validity of Self-Reported Cigarette Smoking in Adults With and Without ADHD. J Dual Diagn. 2019 Jul-Sep;15(3):177-183. doi: 10.1080/15504263.2019.1620399. Epub 2019 Jun 3. PMID 31156069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Smokers and nonsmokers with and without ADHD
Groups:
- Smokers With ADHD: Smokers with ADHD participated in one overnight abstinence condition (withdrawal) and one smoking condition (smoking the first cigarette of the morning).
  Cigarette smoking versus withdrawal in smokers: Each fMRI scan included an experimental task consisting of mathematical problems. Smokers participated in two fMRI scans during the experimental task under the following two conditions: (1) after smoking a cigarette and (2) after overnight abstinence (withdrawal).
- Nonsmokers With ADHD: Nonsmokers with ADHD participated in one fMRI scan during an experimental task consisting of mathematical problems.
- Control Smokers: Control smokers participated in one overnight abstinence condition (withdrawal) and one smoking condition (smoking the first cigarette of the morning).
  Cigarette smoking versus withdrawal in smokers: Each fMRI scan included an experimental task consisting of mathematical problems. Smokers participated in two fMRI scans during the experimental task under the following two conditions: (1) after smoking a cigarette and (2) after overnight abstinence (withdrawal).
- Control Nonsmokers: Control nonsmokers participated in one fMRI scan during an experimental task consisting of mathematical problems.
Period: Overall Study
Arm/Group | Smokers With ADHD | Nonsmokers With ADHD | Control Smokers | Control Nonsmokers
Started | 19 | 21 | 23 | 26
Completed | 19 | 21 | 23 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ADHD Smokers: ADHD smokers participated in two conditions: (1) after smoking a cigarette and (2) after overnight abstinence.
- ADHD Nonsmokers: ADHD nonsmokers participated in the abstinence condition.
- Control Smokers: Control smokers participated in two conditions: (1) after smoking a cigarette and (2) after overnight abstinence.
- Control Nonsmokers: Control nonsmokers participated in the abstinence condition.
- Total: Total of all reporting groups
Arm/Group | ADHD Smokers | ADHD Nonsmokers | Control Smokers | Control Nonsmokers | Total
Number analyzed (Participants) | 19 | 21 | 23 | 26 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.00 (1.70) | 27.24 (7.96) | 25.04 (4.29) | 22.69 (1.85) | 24.44 (4.88)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 6 | 4 | 18 | 30
  Male | 17 | 15 | 19 | 8 | 59
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 23 | 26 | 89

OUTCOME MEASURES:

1. Primary Outcome: Brain Activity
Description: BOLD z-score of smokers with ADHD after abstinence/smoking a cigarette, control smokers after abstinence/smoking a cigarette, nonsmokers with ADHD, and control nonsmokers. All participants performed a mathematical task in the MRI scanner. Higher BOLD z-scores indicate greater brain activation.
Time Frame: One MRI session for nonsmokers and two MRI sessions for smokers
Population: Discrepancies between participant flow and number of participants analyzed are due to motion artifacts, which compromised the MRI findings. Thus, a number of participants had to be excluded from the MRI data analysis.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Smokers With ADHD After Abstinence: Smokers with ADHD after overnight abstinence (withdrawal).
- Nonsmokers With ADHD; Control Nonsmokers: Nonsmokers participate in one condition.
- Control Smokers After Abstinence: Control smokers after overnight abstinence (withdrawal).
- Smokers With ADHD After Smoking: Smokers with ADHD after smoking the first cigarette of the day
- Control Smokers After Smoking: Control smokers after smoking the first cigarette of the day
Arm/Group | Smokers With ADHD After Abstinence | Nonsmokers With ADHD | Control Smokers After Abstinence | Control Nonsmokers | Smokers With ADHD After Smoking | Control Smokers After Smoking
Number analyzed (Participants) | 13 | 14 | 19 | 21 | 13 | 19
z-score
  BOLD Frontal Lobe | 2.08 (0.23) | 2.01 (0.63) | 2.24 (0.18) | 2.30 (0.20) | 2.19 (0.25) | 2.26 (0.23)
  BOLD Parietal Lobe | 2.69 (0.53) | 2.30 (0.37) | 2.48 (0.37) | 2.77 (0.71) | 2.61 (0.72) | 2.60 (0.70)
  BOLD Occipital Lobe | 2.72 (0.47) | 2.87 (0.74) | 2.71 (0.61) | 2.88 (0.49) | 2.80 (0.75) | 2.90 (0.80)
Statistical Analysis 1: Comparison: Smokers With ADHD After Abstinence vs Nonsmokers With ADHD vs Control Smokers After Abstinence vs Control Nonsmokers; Frontal BOLD during abstinence in smokers and nonsmokers; Test type: Superiority or Other; p = 0.46, ANOVA; Threshold for statistical significance p < 0.05; F = 0.56
Statistical Analysis 2: Comparison: Smokers With ADHD After Abstinence vs Nonsmokers With ADHD vs Control Smokers After Abstinence vs Control Nonsmokers; Parietal BOLD during abstinence in smokers and nonsmokers; Test type: Superiority or Other; p = 0.012, ANOVA; Threshold for statistical significance p < 0.05; F = 6.64 — Diagnosis by smoking status interaction
Statistical Analysis 3: Comparison: Smokers With ADHD After Abstinence vs Nonsmokers With ADHD vs Control Smokers After Abstinence vs Control Nonsmokers; Occipital BOLD during abstinence in smokers and nonsmokers; Test type: Superiority or Other; p = 0.04, ANOVA; Threshold for statistical significance p < 0.05; F = 211.20 — Main effect for smoking status
Statistical Analysis 4: Comparison: Smokers With ADHD After Abstinence vs Control Smokers After Abstinence vs Smokers With ADHD After Smoking vs Control Smokers After Smoking; Frontal BOLD smoking versus nonsmoking in smokers with ADHD compared to control smokers; Test type: Superiority or Other; p = 0.22, ANOVA; Threshold for statistical significance p < 0.05; F = 1.6
Statistical Analysis 5: Comparison: Smokers With ADHD After Abstinence vs Control Smokers After Abstinence vs Smokers With ADHD After Smoking vs Control Smokers After Smoking; Parietal BOLD smoking versus nonsmoking in smokers with ADHD compared to control smokers; Test type: Superiority or Other; p = 0.51, ANOVA; Threshold for statistical significance p < 0.05; F = 0.43
Statistical Analysis 6: Comparison: Smokers With ADHD After Abstinence vs Control Smokers After Abstinence vs Smokers With ADHD After Smoking vs Control Smokers After Smoking; Occipital BOLD smoking versus nonsmoking in smokers with ADHD compared to control smokers; Test type: Superiority or Other; p = 0.69, ANOVA; Threshold for statistical significance p < 0.05; F = 0.16

2. Secondary Outcome: DRD4 Genotype
Time Frame: one time blood draw
Population: Discrepancies between participant flow and data analyze reflect that not all participants provided blood samples. Dopamine genotypes were only available for participants who were also enrolled in the Multimodal Treatment for ADHD Study (MTA-Study).
Measure: Count of Participants; unit: Participants
Groups:
- Smokers With ADHD: Smokers with ADHD provided a blood sample.
- Nonsmokers With ADHD: Nonsmokers with ADHD provided a blood sample.
- Control Smokers: Control smokers provided a blood sample.
- Control Nonsmokers: Control nonsmokers provided a blood sample.
Arm/Group | Smokers With ADHD | Nonsmokers With ADHD | Control Smokers | Control Nonsmokers
Number analyzed (Participants) | 10 | 7 | 5 | 18
Participants
  DRD4-4R/7R | 1 | 5 | 2 | 10
  DRD4-4R/4R | 5 | 1 | 3 | 7
  DRD4-3R/4R | 1 | 0 | 0 | 0
  DRD4-3R/3R | 1 | 0 | 0 | 0
  DRD4-2R/4R | 2 | 0 | 0 | 1
  DRD4-2R/2R | 0 | 1 | 0 | 0

3. Secondary Outcome: Salivary Cotinine
Description: Average level of salivary cotinine over all time points (microgram/milliliter)
Time Frame: Once per week for 4 weeks
Population: Discrepancies between participants cotinine samples and participant flow are due to the fact that not all participants provided useful saliva samples.
Measure: Mean (Standard Deviation); unit: Microgram/milliliter
Arm/Group | ADHD Smokers | ADHD Nonsmokers | Control Smokers | Control Nonsmokers
Number analyzed (Participants) | 19 | 14 | 20 | 26
Microgram/milliliter | 100.06 (111.52) | 24.53 (86.66) | 104.99 (84.75) | 23.13 (52.65)

ADVERSE EVENTS:
Time Frame: Up to 6 years.
Groups:
- Control Smokers: Control smokers participated in one overnight abstinence condition (withdrawal) and one smoking condition (smoking the first cigarette of the morning).
  Cigarette smoking versus withdrawal in smokers: Each participant will undergo an fMRI scan during an experimental task consisting of mathematical problems and unpleasant and neutral pictures. Smokers will undergo two fMRI scans during similar experimental tasks under the following two conditions: (1) after smoking a cigarette and (2) after overnight abstinence (withdrawal).
Arm/Group | Smokers With ADHD | Nonsmokers With ADHD | Control Smokers | Control Nonsmokers
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/23 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No